CLINICAL TRIAL: NCT02209649
Title: Bioavailability of Lacidipine 4 mg and Telmisartan 40 mg Administered Orally as Two Experimental Fixed Dose Combination Tablets Relative to Separate Tablets. An Open Randomised Three-way Cross-over Steady State Trial in 6 Female and 6 Male Healthy Subjects
Brief Title: Bioavailability of Lacidipine and Telmisartan Fixed Dose Combination Tablets Relative to Separate Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1173.6
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — lacidipine; Telmisartan; Tablets

ARMS (3):
- Telmisartan and Lacidipine FDC, formulation A (Experimental)
  Interventions: Drug: Lacidipine and Telmisartan fixed dose combination (FDC) tablet
- Telmisartan and Lacidipine FDC, formulation B (Experimental)
  Interventions: Drug: Lacidipine and Telmisartan fixed dose combination (FDC) tablet
- Lacidipine and Telmisartan, mono (Active Comparator)
  Interventions: Drug: Lacidipine; Drug: Telmisartan

INTERVENTIONS:
Drug: Lacidipine and Telmisartan fixed dose combination (FDC) tablet
  Arms: Telmisartan and Lacidipine FDC, formulation A; Telmisartan and Lacidipine FDC, formulation B
Drug: Lacidipine
  Arms: Lacidipine and Telmisartan, mono
Drug: Telmisartan
  Arms: Lacidipine and Telmisartan, mono

SUMMARY:
Study to compare the bioavailability of Lacidipine and Telmisartan administered as fixed dose combination tablets with the separate Telmisartan and Lacidipine tablets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female Caucasian subjects as determined by results of screening
* Age ≥ 18 and ≤ 50 years
* Broca ≥ - 20 % and ≤ + 20 %
* Written informed consent in accordance with Good Clinical Practice and local legislation given

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and electrocardiogram) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Disease of the central nervous system (such as epilepsy) or psychiatric disorders or neurologic disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) (≤ 1 month prior to administration or during the trial, except for oral contraceptives)
* Use of any drugs which might influence the results of the trial (≤ 10 days prior to administration or during the trial except for oral contraceptives)
* Participation in another trial with an investigational drug (≤ 2 months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Blood donation > 100 ml (≤ 4 weeks prior to administration or during the trial)
* Excessive physical activities (≤ 10 days prior to administration or during the trial)
* Any laboratory value outside the reference range of clinical relevance
* Females only:

  * no reliable contraception (e.g. oral contraceptives, 3-month injection, intrauterine device, sterilisation)
  * pregnancy of breast feeding period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 1999-10; Primary Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve at steady state (AUCss) | up to 72 hours after drug administration at day 7
Maximum concentration (Cmax,ss) | up to 72 hours after drug administration at day 7
Time to maximum concentration (tmax) | up to 72 hours after drug administration at day 7
Total apparent clearance (CLtot/f) | up to 72 hours after drug administration at day 7
Apparent volume of distribution (Vz/f) | up to 72 hours after drug administration at day 7
Mean residence time (MRTss) | up to 72 hours after drug administration at day 7
Terminal half-life (t1/2) | up to 72 hours after drug administration at day 7
Number of patients with adverse events | up to 66 days
Number of patients with abnormal findings in physical examination | up to 66 days
Number of patients with clinically relevant changes in electrocardiogram | up to 66 days
Number of patients with clinically relevant changes in vital signs | up to 66 days
Number of patients with abnormal changes in laboratory parameters | up to 66 days
Assessment of tolerability on a verbal rating scale | between day 3 and 5 after last study drug administration